CLINICAL TRIAL: NCT06077214
Title: Liposomal Bupivacaine for Post-operative Pain Control in Adolescent Bariatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20025041
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Bariatric Surgery Candidate; Post-operative Pain
Keywords: liposomal bupivacaine; Exparel
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients will randomly be treated with either liposomal bupivacaine (study drug) or standard bupivacaine after undergoing bariatric surgery.
Who Masked: Participant
Masking Description: Patients will not be told the group to which they were assigned and will have been under anesthesia for administration. The surgeon, other clinical team members, and the study staff will not be blinded to the study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiemental (Experimental): Subjects will be treated with liposomal bupivacaine (study drug) after undergoing bariatric surgery.
  Interventions: Drug: Treatment with liposomal bupivacaine
- Standard of Care (Active Comparator): Subjects will be treated with standard bupivacaine after undergoing bariatric surgery.
  Interventions: Drug: Treatment with standard bupivacaine

INTERVENTIONS:
Drug: Treatment with liposomal bupivacaine — Patients will randomly be treated with either liposomal bupivacaine (study drug) after undergoing bariatric surgery.
  Other Names: Exparel
  Arms: Experiemental
Drug: Treatment with standard bupivacaine — Patients will randomly be treated with standard bupivacaine after undergoing bariatric surgery.
  Arms: Standard of Care

SUMMARY:
Liposomal bupivacaine (trade name Exparel) is a local analgesic that is designed to produce more long-term pain control. Bupivacaine, a widely used local analgesic, is stored within liposomes, which break down in soft tissue over time. Typical length of therapeutic effect for standard bupivacaine is up to 6 hours. The liposomal formulation of bupivacaine, however, has a length of therapeutic effect of up to 72 hours. Typical post-operative incisional pain is known to last for several days in most cases and is thought to peak between 1-2 days after surgery. Therefore, the benefit of most short-acting local analgesics does not overlap with the period of most need.

DETAILED DESCRIPTION:
Use of liposomal bupivacaine has not been reported specifically for use in adolescent bariatric surgery. Our rationale is based on the notion that for most minimally invasive procedures, methods currently used for pain control provide good outcomes that liposomal bupivacaine may not necessarily be able to improve upon. It is critically important to minimize the narcotics for our bariatric surgical patients so they are mobilized early and frequently to minimize their risk for a deep venous thrombosis, which could become a pulmonary embolus. In addition, as these patients are prone to constipation after their operation as a result of their 2 week protein sparing liquid diet preoperatively, avoiding narcotics can reduce their chances of further challenges in return of their bowel function. For these reasons, we seek to investigate whether incorporating liposomal bupivacaine in the analgesic regimen for patients undergoing a laparoscopic sleeve gastrectomy will lead to improvements in patient-reported outcomes and decreased opioid utilization.

ELIGIBILITY:
Inclusion Criteria:

* patients who are undergoing a laparoscopic sleeve gastrectomy for severe obesity who are between 13 and 2018 years of age.
* Only patients treated at the Children's Hospital of Richmond at VCU will be included.

Exclusion Criteria:

* patients less than 13 or greater than 2018 years of age
* patients with an allergy to bupivacaine
* any patients undergoing any additional procedures at the time of the laparoscopic sleeve gastrectomy.
* English or Spanish proficiency will be necessary.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Changed pain scores using liposomal bupivacaine day 1 post-operative | Day 1 post-operative
  Using the 10 point pain scale, determine if liposomal bupivacaine use leads to changed pain scores on post-operative day 1 compared to standard analgesics after laparoscopic sleeve gastrectomy.

SECONDARY OUTCOMES:
Changed pain scores liposomal bupivacaine days 0, 2,3 post-operative | Days 0, 2, 3 post-operative
  Using the 10 point pain scale,determine if liposomal bupivacaine use leads to changed pain scores on post-operative days 0, 2, and 3 compared to standard analgesics after laparoscopic sleeve gastrectomy.
Changed use of opioid medications post operative days 0-3 | Post-operative days 0-3
  To determine if liposomal bupivacaine use leads to changed total consumption of opioid medications after laparoscopic sleeve gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sulkowski, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States